CLINICAL TRIAL: NCT06678438
Title: Brachial Plexus Nerve Block Versus Haematoma Block for Closed Reduction of Distal Radius Fracture in Adults - The BLOCK Trial. A Multicentre Randomised Controlled Trial.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTA no: 2024-512191-35-00
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-11

CONDITIONS: Distal Radius Fractures; Fracture Dislocation; Fracture Dislocation of Upper Limb Joint; Colles' Fracture; Closed Reduction of Fracture and Application of Plaster Cast
Keywords: Lidocaine; Local anaesthesia; Regional anaesthesia; Peripheral nerve block; Brachial plexus block; Lateral infraclavicular block; Axillary plexus block; Distal radius fracture; Colles' fracture; Wrist fracture
MeSH Terms: conditions — Wrist Fractures; Fracture Dislocation; Colles' Fracture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is unfeasible to blind the patients, the doctor who performs the brachial plexus nerve block and the doctor who performs the standard care and the closed reduction. As a result, data on patient evaluated outcomes, i.e. maximum pain score during closed reduction; maximum pain within the first 24 hours after closed reduction; pain at rest; discomfort related to the anaesthetic procedure; overall satisfaction with the treatment; PRWE; DASH; EQ-5D-5L; and data on the closed reduction, i.e. number of attempts used for closed reduction and difficulty of closed reduction of the fracture, will be reported unblinded. Importantly, other caregivers and all outcome assessors are blinded, including the doctor who evaluate the radiographic results and assess the need for surgery, as well as all personnel involved in the subsequent outcome evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Ultrasound-guided brachial plexus nerve block. A total of 30 ml of lidocaine (10 mg/ml) with adrenaline (5 ug/ml) will be administered in multiple injections.
  Interventions: Procedure: Ultrasound-guided brachial plexus block
- Control group (Active Comparator): Haematoma block with local anaesthetics i.e. lidocaine with adrenaline
  Interventions: Procedure: Haematoma Block

INTERVENTIONS:
Procedure: Ultrasound-guided brachial plexus block — The block will be performed as either a lateral infraclavicular brachial plexus block or an axillary brachial plexus block
  Arms: Intervention group
Procedure: Haematoma Block — Participants will receive no peripheral nerve block and receive a haematoma block, with or without supplemental sedation and/or systemic analgesia for the closed reduction according to local guidelines and clinical practices
  Arms: Control group

SUMMARY:
The aim of the project is to evaluate the beneficial and harmful effects of an ultrasound-guided brachial plexus nerve block for patients with a distal radius (wrist) fracture in the need of realignment of fractured bone endings without cutting the skin (closed reduction), in comparison to a haematoma block, which is standard care in Denmark.

Every participant will receive one of the following types of anaesthesia for the realignment of the wrist fracture:

1. A nerve block of the arm (plexus brachialis block)
2. A haematoma block, which is the current standard anaesthesia in the emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years) with a distal radius fracture in need of closed reduction

Exclusion Criteria:

* Patients who would never qualify for surgery according to local guidelines
* Lack of informed consent
* No Danish Central Person Register (CPR) number
* Allergies to the trial medication
* Distal radius fracture initially deemed to require surgery regardless of the outcome of the closed reduction
* Open fractures (fracture-related wound requiring sutures)
* Other fractures on the same extremity ((NOT including distal ulna fracture(s))
* Bilateral distal radius fractures both requiring closed reduction
* Concomitant medical or surgical condition taking priority over the closed reduction of the distal radius fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1716 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative proportion of patients with distal radius fracture surgery | 90 days after closed reduction

SECONDARY OUTCOMES:
Composite outcome of treatment related complications | 90 days after closed reduction
  loco-regional neurological complications from affected arm, local anaesthetic systemic toxicity, soft tissue injuries (including skin injuries) related to the closed reduction procedure, infection at the site of needle puncture, vessel puncture requiring subsequent treatment (including compression), pneumothorax, allergic reaction, new bone or joint injury (e.g. dislocation or fracture) after the closed reduction and/or pulmonary embolism
Patient Rated Wrist Evaluation (PRWE) | 90 days after closed reduction
  The PRWE is a patient-reported outcome and the PRWE-score is calculated from the Danish-validated translation of the PRWE questionnaire
Maximum pain score in the affected wrist during closed reduction(s) | 0-12 hours after the closed reduction
  The pain outcomes are patient-reported as a Numerical Rating Scale (NRS) score on a scale from 0=no pain to 10=worst pain imaginable. If the patient has the closed reduction performed more than one time, the patient will be asked to report the worst pain experienced during all the attempts of a closed reduction.
Proportion of patients with unacceptable radiographic fracture position immediately after closed reduction | 0 -24 hours after closed reduction
  The radiographic fracture position is evaluated according to the American Academy of Orthopaedic Surgerons (AAOS) guidelines. The fracture position is unacceptable if the fracture has a radial shortening > 3 mm, > 10 degrees dorsal tilt of the articular surface of radius from a perpendicular line on the longitudianal axis of radius or intra-articular displacement or step-off > 2 mm.

OTHER OUTCOMES:
Pain at rest in the affected wrist immediately, 90 days, and 12 months after closed reduction | 0-12 hours, 90 days and 12 months after closed reduction
  The pain outcomes are patient-reported as a Numerical Rating Scale (NRS) score on a scale from 0=no pain to 10=worst pain imaginable.
Maximum pain in the affected wrist within the first 24 hours after closed reduction | 24-36 hours after the closed reduction.
  The pain outcomes are patient-reported as an NRS score on a scale from 0=no pain to 10=worst pain imaginable.
Proportion of patients with complex regional pain syndrome (CRPS) | 90 days and 12 months after closed reduction
  CRPS is defined according to the Budapest Criteria
Disabilities of the Arm, Shoulder, and Hand (DASH) score | 90 days and 12 months after closed reduction
  DASH-score is calculated from the Danish-validated translation of the DASH questionnaire
Patient Rated Wrist Evaluation (PRWE) | 12 months after closed reduction
  PRWE-score is calculated from the Danish-validated translation of the PRWE questionnaire
Quality of life (EQ-5D-5L) score | 90 days and 12 months after closed reduction
  The Danish translation of the EQ-5D-5L questionnaire is used and the EQ-5D-5L-score is calculated based on the Danish EQ-5D-5L value set
Number of attempts used for closed reduction | Immediately after closed reduction
Difficulty of closed reduction of the fracture | Immediately after closed reduction
  The doctor reported ease on a numeric rating scale from 0-10; 0=very easy, 10=very difficult)
Discomfort related to the anaesthetic procedure | 0-12 hours after closed reduction
  The discomfort is a patient-reported outcome on a numeric rating scale from 0-10; 0=no discomfort, 10=very uncomfortable
Overall satisfaction with the treatment 0 to 24 hours after initiation of the anaesthesia | 24 hours after closed reduction
  The overall satisfaction is a patient-reported outcome on a numeric rating scale from 0-10; 0=very unsatisfied, 10=very satisfied. When evaluating the treatment, the patient is specifically asked to include all elements of the treatment including: the anaesthetic (procedure and following effects), the experience during the closed reduction and the pain and general sensation in the arm/wrist in the first 24 hours after the treatment commencement.
Proportion of patients with unacceptable radiographic position at first follow-up in the orthopaedic out-patient clinic (typically 10-14 days post-reduction) | 10-14 days after closed reduction
  The radiographic fracture position is evaluated according to the American Academy of Orthopaedic Surgerons (AAOS) guidelines. The fracture position is unacceptable if the fracture has a radial shortening > 3 mm, > 10 degrees dorsal tilt of the articular surface of radius from a perpendicular line on the longitudianal axis of radius or intra-articular displacement or step-off > 2 mm.
Proportion of individual complications in the composite secondary outcome | 90 days after closed reduction
Proportion of patients having one or more serious adverse events (SAEs), including events related to loss of hand function | Within 90 days after closed reduction
  A SAE is defined as an adverse event that leads to the following incidents:
  * Death
  * Life threatening injury or disease
  * Severe or permanent disability
  * Admission to the hospital or prolongation of hospitalisation
  Surgical reduction of the distal radius fracture, including relevant admission to hospital, will not be catagorised as a SAE.
Proportion of patients having one or more adverse events (AEs) | Within 24 hours after closed reduction
  An AE is defined as any harmful and unintended event, sign, or symptom, that appear during the trial period, regardless of whether this AE is considered related to the treatment or not.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie D Harwood, MD, PhD-fellow, Principal Investigator — Copenhagen University Hospital - North Zealand; Anne-Sofie Jellestad, MD, PhD-fellow, Principal Investigator — Copenhagen University Hospital - North Zealand
Locations (1):
- Copenhagen University Hospital - North Zealand Hillerød, Hillerød, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupont Harwood C, Jellestad AL, Bahuet AR, Knudsen RL, Andersen LC, Mathiesen O, Asko Andersen J, Jakobsen JC, Rothe C, Jorgensen CC, Viberg B, Brorson S, Brabrand M, Gundtoft PH, Terndrup M, Lange KHW, Lundstrom LH, Norskov AK. Brachial plexus nerve block versus haematoma block for closed reduction of distal radius fracture in adults: The BLOCK Trial - a protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Jul 8;15(7):e099954. doi: 10.1136/bmjopen-2025-099954. PMID 40633950